CLINICAL TRIAL: NCT00893906
Title: Assessment of the Effectiveness of Seasonal Trivalent Influenza Vaccine Among Children in Senegal
Brief Title: Inactivated Influenza Vaccine Effectiveness in Tropical Africa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Institut de Recherche pour le Developpement (Other Government); Institut Pasteur (Industry); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TIV-SEN-01
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Influenza
Keywords: influenza; influenza vaccine; vaccine effectiveness; cluster randomized; Africa
MeSH Terms: conditions — Influenza, Human | interventions — vaxigrip; Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIV (Experimental): Children living in villages randomized to influenza vaccine
  Interventions: Biological: seasonal trivalent inactivated influenza vaccine
- IPV (Experimental): Children living in villages randomized to polio vaccine
  Interventions: Biological: inactivated polio vaccine

INTERVENTIONS:
Biological: seasonal trivalent inactivated influenza vaccine — vaccine to be used according to marketed dosage and frequency
  Other Names: Vaxigrip
  Arms: TIV
Biological: inactivated polio vaccine — vaccine to be used according to marketed dosage and frequency
  Other Names: Imovax Polio
  Arms: IPV

SUMMARY:
Influenza, a highly communicable acute respiratory disease, is one of the major infectious disease threats to the human population. In Africa, information on the occurrence of influenza and its disease burden is seriously lacking. Such data would be important in determining the contribution of influenza to the more than two million annual pneumonia deaths among children globally, mostly in the developing world, and the potential number of deaths that could be prevented by influenza vaccination.

A single dose of trivalent inactivated influenza vaccine (TIV) is 70 to 90 percent effective in preventing influenza in healthy older children and young and middle-aged adults, but is less efficacious in young children and the elderly. Young children who suffer substantial influenza morbidity and are unlikely to have pre-existing immunity should receive two doses of TIV to provide adequate immunity. Because family studies of influenza transmission conducted during the 1970's found children to be the main introducers of influenza into households, vaccination of children may decrease the chances of spreading influenza to contacts. Mass vaccination of schoolchildren has been correlated with reduced respiratory illness in unvaccinated persons suggesting that immunization of children on a larger scale can affect community epidemics.

In temperate industrialized countries with seasonal disease, influenza vaccine is given annually, prior to the influenza season, and generally targeted to individuals with the highest risk of severe disease. Influenza prevention strategies may need to differ in tropical developing countries due to a variety of reasons. Given the varying influenza circulation patterns, it is unknown which hemisphere vaccine formulation will provide year-round protection against the diverse strains that may exist in tropical countries. Persons residing in developing countries also may have nutritional deficiencies or underlying diseases and infections that affect vaccine immunogenicity. Consideration must be given to programmatic issues as well. Adolescent and adult preventive health services are poorly developed in many countries, and thus a strategy that targets children may be the most feasible option. In addition, vaccinating children may be the most cost-effective option, as it has the potential to provide direct benefit to those vaccinated, as well as indirect benefits to unvaccinated members of the population. Thus, an influenza vaccine effectiveness study in a tropical developing country population will help to elucidate burden of seasonal influenza and may inform optimal use of vaccine for either seasonal and pandemic situations.

Thus, this study in Senegal will to evaluate the direct effects of TIV in reducing the occurrence of laboratory-confirmed influenza among children who receive it as well as the potential indirect effects experienced by the population as a result of reducing transmission among children.

DETAILED DESCRIPTION:
The trial will take place in the study area of the Niakhar demographic surveillance system in Senegal, a population representative of rural impoverished Africa. Villages will be randomized to TIV or a beneficial control vaccine-inactivated polio vaccine-and children 6 months to 10 years of age will be targeted for vaccination. Four hundred children will be further enrolled into an immunogenicity and safety substudy which will measure their immune response to vaccination and assess in detail reactions and adverse events to the vaccines in these populations. For evaluation of effectiveness, passive and active surveillance will be conducted to identify laboratory-confirmed influenza among enrolled children and in the population in which they live. Such surveillance will also allow a determination of the rates of influenza and a description of the clinical characteristics of the disease in an African population. With such epidemiologic data, national and global public health officials will have better data for developing future influenza control strategies for either seasonal or pandemic influenza.

ELIGIBILITY:
Inclusion Criteria:

* A male or female child at least 6 months of age and no older than 10 years of age (has not yet reached 11 years of age) at the enrollment visit.
* A child whose parent or guardian's primary residence, at the time of study vaccinations, is a village compound selected to receive TIV or IPV.
* Subject's parent or legal guardian is willing to provide written informed consent prior to the subject's first study vaccination.

Exclusion Criteria:

* Hypersensitivity to the active substance or any component in either TIV (which includes egg protein) or IPV. (Please see information on composition of vaccines.)
* Hypersensitivity after previous administration of any influenza or polio vaccine.
* Acute severe febrile illness. (Administration of TIV or IPV should be postponed until after recovery. Minor illnesses, such as mild upper respiratory infection, with or without low grade fever, are not reason for postponing vaccination. Acute severe febrile illness is only a temporary exclusion.)
* Any condition that, in the opinion of the investigator, would pose a health risk to the participant or interfere with the evaluation of the study objectives.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10000 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Total effectiveness of vaccine against laboratory-confirmed symptomatic influenza. | Two weeks post-vaccination through February 28 the following calendar year

SECONDARY OUTCOMES:
Indirect effectiveness against laboratory-confirmed symptomatic influenza | Two weeks post-vaccination through February 28 the following calendar year
Overall effectiveness of vaccine against laboratory-confirmed symptomatic influenza | Two weeks post-vaccination through February 28 the following calendar year
Direct effectiveness of vaccine against laboratory-confirmed symptomatic influenza | Two weeks post-vaccination through February 28 the following calendar year

CONTACTS AND LOCATIONS:
Overall Officials: John C Victor, PhD, MPH, Study Director — PATH; Aldiouma Diallo, MD, Principal Investigator — IRD
Locations (1):
- Niakhar Demographic Surveillance System, Niakhar, Fatick District, Senegal

REFERENCES:
- [Derived] Niang MN, Sugimoto JD, Diallo A, Diarra B, Ortiz JR, Lewis KDC, Lafond KE, Halloran ME, Widdowson MA, Neuzil KM, Victor JC. Estimates of Inactivated Influenza Vaccine Effectiveness Among Children in Senegal: Results From 2 Consecutive Cluster-Randomized Controlled Trials in 2010 and 2011. Clin Infect Dis. 2021 Jun 15;72(12):e959-e969. doi: 10.1093/cid/ciaa1689. PMID 33165566
- [Derived] Diallo A, Diop OM, Diop D, Niang MN, Sugimoto JD, Ortiz JR, Faye EHA, Diarra B, Goudiaby D, Lewis KDC, Emery SL, Zangeneh SZ, Lafond KE, Sokhna C, Halloran ME, Widdowson MA, Neuzil KM, Victor JC. Effectiveness of Seasonal Influenza Vaccination in Children in Senegal During a Year of Vaccine Mismatch: A Cluster-randomized Trial. Clin Infect Dis. 2019 Oct 30;69(10):1780-1788. doi: 10.1093/cid/ciz066. PMID 30689757